CLINICAL TRIAL: NCT00440934
Title: Étude de Phase II Pour déterminer l'efficacité Des Ondes électromagnétiques de Basse intensité administrées Par Voie Buccale Dans le Traitement du Cancer du Foie avancé
Brief Title: A Study of Electromagnetic Waves in the Treatment of the Advanced Hepatocarcinoma
Acronym: THBC002
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor patient accrual
Sponsor: Pasche, Boris, M.D. (Individual)
Collaborators: Barbault, Alexandre, M.S. (Individual)
Responsible Party: Boris Pasche, Boris Pasche
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THBC 002
Record Dates: First submitted 2007-02-24; First posted 2007-02-27 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-05

CONDITIONS: Carcinoma, Hepatocellular
Keywords: carcinoma, hepatocellular; electromagnetic fields
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Amplitude-modulated electromagnetic fields

SUMMARY:
Hepatocarcinoma (HCC) is the first cause of deaths due to cancer worldwide. More than one million two hundred thousand new patients are diagnosed each year. The prognosis of patients suffering from advanced hepatocarcinoma is poor with an average survival of less than six months. Phase I data suggest that low levels of electromagnetic fields administered intrabucally with a portable and programmable device are a safe and potentially effective treatment for advanced cancer. The device is connected to a spoon-like coupler placed in the patient's mouth during treatment. Patients with advanced HCC and limited therapeutic options will be offered treatment with a combination of frequencies.

DETAILED DESCRIPTION:
Hepatocarcinoma (HCC) is the first cause of deaths due to cancer worldwide. More than one million two hundred thousand new patients are diagnosed each year. The prognosis of patients suffering from advanced hepatocarcinoma is poor with an average survival of less than six months. Therapies for hepatocarcinoma are limited. Resection of the primary tumor is the therapeutic approach of first choice when possible. Although this intervention results in long-term survival for some patients, only a minority of them are surgical candidates because of limitations due to tumor size, patient's overall condition or presence of hepatic cirrhosis.

Phase I data suggest that low levels of amplitude-modulated electromagnetic fields administered intrabucally with a portable and programmable device are a safe and potentially effective treatment for advanced cancer. The device is connected to a spoon-like coupler placed in the patient's mouth during treatment. Patients with advanced HCC and limited therapeutic options will be offered treatment with a combination of HCC-specific frequencies.

The patients will be offered ambulatory treatment, which will be administered three times a day for 60 min until disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

* The patients must have a diagnosis of inoperable hepatocellular carcinoma.
* The patients who have an AFP level higher than 400 ng/ml and an appearance characteristic of cancer of the liver do not need histological confirmation. These patients must however have a negative serology for the antigen of surface of hepatitis B If serology for this antigen is positive, they must have a rate of AFP higher than 4000 ng/ml.
* Presence of one or more lesions measurable(s) according to criteria's RECIST.

Exclusion Criteria:

* Other anti-cancer treatments are not authorized during this study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Estimated); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
• To determine disease free survival at 4 months while receiving the experimental treatment. | 4 months
Response rate | six months

SECONDARY OUTCOMES:
To determine the influence of the treatment on the hepatic function of patients with a diagnosis of cirrhosis. To determine the impact of the treatment by means of electromagnetic waves on the overall survival of patients. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Boris Pasche, MD, PhD, Principal Investigator — Cabinet Médical Avenue de la gare 6
Locations (1):
- Cabinet Médical de l'Avenue de la gare 6, Lausanne, Canton of Vaud, Switzerland